CLINICAL TRIAL: NCT05797402
Title: Construction of Integrated Management and Sharing Platform for Clinical and Biological Sample Database of Chinese Elderly Patients With Multiple Diseases
Brief Title: Clinical and Biological Sample Database of Chinese Elderly Patients With Multiple Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Tiantan Hospital (Other); Beijing Geriatric Hospital (Other); China-Japan Friendship Hospital (Other); Xuanwu Hospital, Beijing (Other); Wuhan TongJi Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine,Director,Department of Cardiology, Beijing Anzhen Hospital
Other Study IDs: 2020YFC2004800
Record Dates: First submitted 2023-02-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Comorbidities and Coexisting Conditions; Old Age; Debility
Keywords: Cognition Disorders; Frailty; Coronary heart disease; Atrial fibrillation; Stroke; Heart failure; Hypertension; Valvular heart disease
MeSH Terms: conditions — Frailty; Cognition Disorders; Coronary Disease; Atrial Fibrillation; Stroke; Heart Failure; Hypertension; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- young-aged patients: Patients aged 18 to 45 years old.
- middle-aged patients: Patients aged 46 to 64 years old.
- elderly patients: Patients aged 65 and older.

SUMMARY:
The investigators aim to establish a clinical database and biobank for elderly patients with multiple diseases. The collected data will include demographic information, comorbidity characteristic, FRAIL scale, age-adjusted Charlson comorbidity index, relevant blood tests, the results of imaging examination, prescription of drugs, length of hospital stay, number of overall rehospitalizations and death. With this database, the investigators intend to formulate an individualized treatment strategy for these patients.

DETAILED DESCRIPTION:
According to the China Health and Aging Tracking Survey, a significant proportion of elderly individuals aged over 65 suffer from two or more chronic diseases, with prevalence rates ranging from 22.5% to 47.5%. However, due to the decentralized storage of health data, lack of standardization, and collaboration barriers, it is challenging to make use of this information in a meaningful way.Therefore, there is an urgent need to overcome the technical challenges and build an intelligent diagnosis and treatment system for this vulnerable population.

To achieve this goal, it is necessary to establish a clinical database and biobank that includes data on all elderly patients with multimorbidity. This will enable researchers to conduct clinical research on various factors, including clinical and biological predictors of adverse events such as emergency visits, strokes, heart failure, myocardial infarction, tumors, and acute chronic obstructive pulmonary disease. Additionally, the database will facilitate the development of systematic and individualized evaluation tools for elderly patients with multimorbidity, identify prognostic factors that improve short- and long-term outcomes, and enable the participation in multi-center trials at the national or international level. Ultimately, this effort will help establish clinical database and biobank data collection standards for future studies.

ELIGIBILITY:
Inclusion Criteria:

* (1) written and informed consent, (2) participants aged 18 years or older.

Exclusion Criteria:

* (1) Unwilling to participate in the study, (2) Unable or unwilling to cooperate with the baseline or follow-up data collection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of geriatric syndromes including falls, cognitive impairment, dizziness and frailty | 1 year
  collection of clinical data in the medical record and follow-up update

SECONDARY OUTCOMES:
The incidence of survival rate | 1 year
  collection of clinical data in the medical record and follow-up update

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang X, Zheng W, Wang X, Suo M, Zhao X, Nie S. Association between Charlson Comorbidity Index and in-hospital outcomes among aortic stenosis patients undergoing aortic valve replacement: an observational study at the National Clinical Research Center for Cardiovascular Diseases. BMJ Open. 2025 Jun 17;15(6):e083677. doi: 10.1136/bmjopen-2023-083677. PMID 40527568
- [Derived] Zheng W, Huang X, Wang X, Suo M, Yan Y, Gong W, Ai H, Que B, Nie S. Impact of multimorbidity patterns on outcomes and treatment in patients with coronary artery disease. Eur Heart J Open. 2024 Mar 27;4(2):oeae009. doi: 10.1093/ehjopen/oeae009. eCollection 2024 Mar. PMID 38544919